CLINICAL TRIAL: NCT02623816
Title: Prospective Study Assessing Patient Satisfaction of Symptom Control With Proton Pump Inhibitor Dosing Regimen
Brief Title: Symptom Control Satisfaction With Proton Pump Inhibitor Regimen
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: MetroHealth Medical Center (Other)
Responsible Party: Principal Investigator, Nisheet Waghray, Investigator, MetroHealth Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB13-00089
Record Dates: First submitted 2015-11-29; First posted 2015-12-08 (Estimated); Results first posted 2022-10-25 (Actual); Last update posted 2022-10-25 (Actual); Status verified 2022-10

CONDITIONS: Heartburn
MeSH Terms: conditions — Heartburn | interventions — Omeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sub-optimal dosing (No Intervention): No change will be made to the sub-optimal dosing regimen of omeprazole 20 mg. Rescue antacid use is permitted. Total duration of 6 weeks.
- Optimal dosing (Experimental): Patients will be administered optimal dosing regimen of Omeprazole 20 mg for 4 weeks starting at week 2. Rescue antacid use is permitted. Total duration of 6 weeks.
  Interventions: Drug: Optimal Dosing of Omeprazole

INTERVENTIONS:
Drug: Optimal Dosing of Omeprazole — Omeprazole 20 mg
  Other Names: omeprazole
  Arms: Optimal dosing

SUMMARY:
The overall aim of this study is to assess if patients with persistent gastroesophageal reflux disease (GERD) symptoms receiving sub-optimal omeprazole dosing experience improvement in GERD symptoms when prescribed an optimal dosing regimen. The optimal dosing regimen is defined as taking omeprazole 30 minutes prior to the first meal of the day.

DETAILED DESCRIPTION:
GERD remains a common gastrointestinal complaint, resulting in 6% of outpatient visits. The economic burden is significant with direct costs exceeding $12 billion/year and indirect cost as high as $75 billion/year. The primary aim of this study was determine whether a brief educational intervention optimizing proton pump inhibitor (PPI) dosing would reduce GERD symptoms using the gastroesophageal reflux disease symptom assessment scale (GSAS) questionnaire. Further, secondary analysis would utilize the results of the trial and combine them with costs related to uncontrolled GERD to estimated the potential economic impact.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old
* taking omeprazole 20 mg
* episodic heartburn at least 3 times per week
* provides consent and be willing to complete study questionnaires
* read, speak and write English

Exclusion Criteria:

* weight loss (alarm symptom)
* normal esophagogastroduodenoscopy (EGD) in last one year
* pregnant or women planning on becoming pregnant at any time during the study
* history of Barrett's esophagus
* prior esophageal strictures
* intolerance/allergy to study medications
* patients on plavix or a history of upper gastrointestinal surgery
* investigators or their immediate family (spouse, children, sibling)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2014-08; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: M. Michael Wolfe, MD, Principal Investigator — MetroHealth Medical System
Locations (1):
- MetroHealth Medical System, Cleveland, Ohio, United States

REFERENCES:
- [Result] Waghray A, Waghray N, Perzynski AT, Votruba M, Wolfe MM. Optimal Omeprazole Dosing and Symptom Control: A Randomized Controlled Trial (OSCAR Trial). Dig Dis Sci. 2019 Jan;64(1):158-166. doi: 10.1007/s10620-018-5235-9. Epub 2018 Aug 9. PMID 30094626

RESULTS

PARTICIPANT FLOW:
Groups:
- Sub-optimal Dosing: No change will be made to the sub-optimal dosing regimen of omeprazole 20 mg. Rescue antacid use is permitted. Total duration of 10 weeks.
- Optimal Dosing: Patients will be administered optimal dosing of Omeprazole 20 mg for 4 weeks starting at week 2. Rescue antacid use is permitted. Total duration of 6 weeks.
  Optimal Dosing of Omeprazole: Omeprazole 20 mg
Period: Overall Study
Arm/Group | Sub-optimal Dosing | Optimal Dosing
Started | 40 | 24
Completed | 38 (Two subjects discontinued participation.) | 22
Not Completed | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Optimal Dosing: Patients will be administered optimal regimen dosing of Omeprazole 20 mg for 4 weeks starting at week 2. Rescue antacid use is permitted. Total duration of 6 weeks.
  Optimal Dosing of Omeprazole: Omeprazole 20 mg
- Total: Total of all reporting groups
Arm/Group | Sub-optimal Dosing | Optimal Dosing | Total
Number analyzed (Participants) | 40 | 24 | 64
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.9 (12.2) | 52.3 (13.4) | 51.1 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 15 | 38
  Male | 17 | 9 | 26
Region of Enrollment [Number; unit: Participants]
  United States | 40 | 24 | 64

OUTCOME MEASURES:

1. Primary Outcome: Symptom Frequency and Severity/Distress Scores From Gastroesophageal Reflux Disease Symptom Assessment Scale (GSAS) (Overall)
Description: The 15-symptom GSAS questionnaire includes measures of: Gastrointestinal distress, Regurgitation/heartburn and Upper respiratory manifestations. The outcome measures were the number, frequency, and severity of GSAS symptoms reported at 6 weeks. Measures were based on aggregate GSAS scores. Symptom numbers range from 0 to 15. Frequency is based on the total number of reported days of symptomatic episodes in the past week divided by the number of potential symptoms (number reported divided by 15 for GSAS score. The range for frequency score:0 to 7 with higher scores indicative of greater frequency of symptoms. Severity is the average distress score reported by individuals (zero if no symptoms). Symptom distress is based on a 4 point Likert scale (0= not at all, 1=somewhat, 2=quite a bit and 3=very much). The higher the score the worse outcome.
  .
Time Frame: 6 weeks
Measure: Mean (Standard Error); unit: score on a scale
Groups:
- Sub-optimal Dosing: Continue Current PPI Dosing
- Optimal Dosing: Continue Current Optimal PPI dosing
Arm/Group | Sub-optimal Dosing | Optimal Dosing
Number analyzed (Participants) | 40 | 24
score on a scale
  GSAS Symptoms Score | 8.5 (0.7) | 5.2 (0.5)
  GSAS Frequency Score | 2.2 (0.3) | 1.0 (0.2)
  GSAS Severity Score | 1.0 (0.1) | 0.6 (0.1)

ADVERSE EVENTS:
Time Frame: Adverse event and/or serious adverse event data were collected for 1 year after study enrollment for each study participant.
Arm/Group | Sub-optimal Dosing | Optimal Dosing
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/24
Other Adverse Events (participants affected / at risk) | 0/40 | 0/24

LIMITATIONS AND CAVEATS:
1. Single healthcare system
2. Symptom scoring questionnaire
3. Study did not assess gastric pH

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No